CLINICAL TRIAL: NCT07146191
Title: A Phase 1, Open-label, Single Period Study to Evaluate the Absorption, Metabolism, and Excretion of a Single Microdose of [14C]-RE104 in Healthy Participants
Brief Title: RE104 Radiolabeled Mass Balance (hAME) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reunion Neuroscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE104-103-NHV
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participant Study
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 30 mg 2-[14C]-RE104 (1uCi/30mg) (Experimental): A single subcutaneous injection of 30 mg 2-[14C]-RE104 for Injection
  Interventions: Drug: 2-[14C]-RE104 for Injection

INTERVENTIONS:
Drug: 2-[14C]-RE104 for Injection — Single, subcutaneous dose of 2-[14C]-RE104 for Injection

SUMMARY:
The purpose of this study is to characterize the absorption, metabolism and routes of excretion of RE104 and its metabolites in healthy volunteers. This study will quantify drug and metabolites in blood, urine, and feces samples collected before study drug administration and through at least 168 hours after SC dosing of [14C]-RE104.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age (inclusive), and a body mass index of 18-34 kg/m2.
* Willing to take a drug with psychoactive properties
* If female and of childbearing potential, agrees to use an acceptable method of birth control and is not planning to become pregnant before, during or within 90 days after the last dose of the study drug.
* If male, must agree to use condom with spermicide during and up to 90 days after discharge."
* Must agree to refrain from sperm or egg donation until 120 days post discharge.
* Able to understand and adhere to study schedule and requirements and willing to sign an ICF
* In good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening
* Agrees to not participate in other research studies involving investigational medication or medical devices for the duration of the study

Exclusion Criteria:

* Active or medical history of bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorder and/or borderline personality disorder, or first-degree family history of psychosis or bipolar disorder.
* Medical condition or other concomitant condition or history rendering unsuitability for the study
* Has used or intends to use prohibited medications
* Has a known sensitivity or intolerance to hallucinogenic or psychedelic substances, or potential rescue medications
* Has participated in another clinical study within 30 days and/or with a [14C] labeled study drug within 1 year prior to enrolling.
* Is pregnant or has a female partner who is pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Total excreted radioactivity (Ae) | Through 168 hours postdose
Cumulative recovery of total excreted radioactivity (CUM Ae) | Through 168 hours postdose
Area under the concentration-time curve (AUC) for RE104 and 4-OH-DiPT | Through 168 hours postdose
Maximum observed concentration (Cmax) for RE104 and 4-OH-DiPT | Through 168 hours postdose
Time to reach Cmax (Tmax) for RE104 and 4-OH-DiPT | Through 168 hours postdose
Terminal half-life (t1/2) of RE104 and 4-OH-DiPT | Through 168 hours postdose
Apparent terminal elimination half-life (λz) for RE104 and 4-OH-DiPT | Through 168 hours postdose
Mean residence time (MRT) | Through 168 hours postdose
Apparent total body clearance (CL/F) for RE104 | Through 168 hours postdose
Apparent volume of distribution during the terminal phase (Vz/F) for RE104 | Through 168 hours postdose
Total metabolite profiling with description of relevant PK parameters and structural identification of major metabolites present in all matrices | Through 168 hours postdose

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) by frequency, severity and seriousness | From dosing (Day 0) through study completion (Day 7)
  A treatment-emergent adverse event (TEAE) is defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, Chief Medical Officer, Study Director — Reunion Neuroscience Inc
Locations (1):
- PPD Inc., Austin, Texas, United States